CLINICAL TRIAL: NCT04219215
Title: Acute Hyperbaric Oxygen (HBO) Treatment Increases Hepatic Insulin Sensitivity and Muscle Reactive Oxygen Species in Type 2 Diabetes
Brief Title: Acute Hyperbaric Oxygen Treatment Increases Hepatic Insulin Sensitivity and Muscle Reactive Oxygen Species in T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HBO
Record Dates: First submitted 2019-09-11; First posted 2020-01-06 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Type 2-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygenation (Experimental): Patients with T2D receive an 2 hour treatment with 100 % oxygen in a hyperbaric chamber
  Interventions: Device: 100% O2 in oxygen chamber; Device: 21% O2 in oxygen chamber
- Ambient Air (Experimental): Patients with T2D receive an 2 hour treatment with 21% oxygen in a hyperbaric chamber
  Interventions: Device: 100% O2 in oxygen chamber; Device: 21% O2 in oxygen chamber

INTERVENTIONS:
Device: 100% O2 in oxygen chamber — Application of 100% O2 in an hyperbaric oxygen chamber
Device: 21% O2 in oxygen chamber — Application of ambient air (21% O2) in an hyperbaric oxygen chamber

SUMMARY:
Diabetes mellitus type 2 (T2D) is characterized by insulin resistance of liver and skeletal muscle, which is at least partly due to impaired muscle mitochondrial function. Long-term HBO therapy, as applied for treating the diabetic foot syndrome, has been shown to improve blood glucose concentrations. To study the underlying mechanisms, we want to examin the short-term effect of HBO treatment on insulin sensitivity and mitochondrial oxidative capacity and production of reactive oxygen species (ROS) in a randomized, double blinded, placebo-controlled cross-over trial.

DETAILED DESCRIPTION:
In total 14 patients are planned. Each participant participates in both experimental parts (100% O2 and ambient air). They are examined immediately after each HBO/ ambient air therapy. The allocation is randomized treated every three weeks with 2-hour therapies using pure O2 or indoor air. Randomized and double-blinded in a cross-over setting, one group of patients with type 2 diabetes is first treated with HBO therapy and the other group is first treated with room air. Here, an ambient pressure of 2.4 ATM is built up and then administered for respiration over a total of 90 minutes of pure O2. Patients are examined on two consecutive days for each part of the study.On the first day serum samples are taken and a sample is taken from the vastus lateralis muscle. A magnetic resonance spectroscopic examination (MRS) is performed on the patient subsequently. In this case, phosphorus metabolites (absolute quantification of ATP, Pi) and the ATP synthase flow rate (fATP) are determined non-invasively by means of 31P MRS and TG storage (HCL) by means of 1H-MRS.

On the next day of the trial patients are treated with HBO therapy or room air. A hyperinsulinemic-euglycemic clamp test (120-300 min) with administration of deuterated glucose (D- [6,6-2H2] glucose) (0-120 min) to measure muscular and hepatic insulin resistance will be performed after the end of HBO therapy or room air treatment performed. Indirect calorimetry determines energy consumption and substrate selection (lipid and glucose oxidation) in hyperinsulinaemia. After the end of the HBO therapy or room air treatment and 30 minutes after the start of the clamp test, a sample is taken from the vastus lateralis muscle again.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years
* Type 2 diabetes
* HbA1c ≥ 6 and ≤ 9%
* BMI ≤ 35 kg / m2

Exclusion Criteria:

* Treatment with thiazolidinedione in the last 6 months
* Uncontrolled hyperglycemia (FPG ≥ 240 mg / dl)
* vitamin supplement (washing out at least 4 weeks)
* Patients requiring revascularization
* Serum CRP ≥ 5 mg / dl
* Previous treatment for HBO therapy
* Secondary diabets according to ADA criteria (type 3 B-H, eg pancreopriver diabetes)
* Type 4 diabetes (gestational diabetes), pregnancy
* poor glycemic control (HbA1c> 9.0%)
* Hyperlipidemia (low density triglycerides and lipoproteins ≥ double upper Reference limit)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Change in rate of glucose disappearance | 12 months
  measurement of whole body insulin sensitivity with hyperinsulinamic euglycemic clamp test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarabhai T, Mastrototaro L, Kahl S, Bonhof GJ, Jonuscheit M, Bobrov P, Katsuyama H, Guthoff R, Wolkersdorfer M, Herder C, Meuth SG, Dreyer S, Roden M. Hyperbaric oxygen rapidly improves tissue-specific insulin sensitivity and mitochondrial capacity in humans with type 2 diabetes: a randomised placebo-controlled crossover trial. Diabetologia. 2023 Jan;66(1):57-69. doi: 10.1007/s00125-022-05797-0. Epub 2022 Sep 30. PMID 36178534